CLINICAL TRIAL: NCT00201474
Title: Signs of Organic Brain Dysfunction in Psychiatric Patients With Fluctuating Psychiatric Symptoms Including Brief Depressions Compared to Patients With a Major Depressive Episode.
Brief Title: Acute, Affective, Organic Disorders.
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Dr. Dedichens Institute for Psychiatric Research, Oslo, Norway. (Unknown); GlaxoSmithKline (Industry)
Responsible Party: Prof Olav Linaker, St Olavs University Hospital, Division Psychiatry, Norwegian University of Science and Technology
Other Study IDs: AEV-98
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Depressive Disorders
Keywords: brief depressive episodes; affective disorders; EEG and QEEG; epilepsy; organic brain disorders; acute psychiatry
MeSH Terms: conditions — Depressive Disorder; Mood Disorders; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Ordinary laboratory tests, medication, substances.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- brief depressive periods: brief depressive periods together with other fluctuating psychiatric symptoms
- major depressive disorder

SUMMARY:
The purpose of the study is to investigate whether patients with brief depressive periods together with other fluctuating psychiatric symptoms, have this condition due to epilepsy or an other organic brain disorder.

DETAILED DESCRIPTION:
A limited number of patients admitted to psychiatric acute wards or Psychiatric Intensive Care Units are admitted with a fluctuating array of psychiatric symptoms including brief depressive episodes. These patients do not fit into the present diagnostic systems due to short duration of affective symptoms and the fluctuating arrays of other symptoms. Case histories indicate that these patients have psychiatric conditions due to epilepsy or organic brain dysfunctions.

In the study acutely admitted patients filling criteria for two recent DSM-4 axis 1 diagnoses (one is a brief depressive period) during the last two weeks are compared to age- and sex-matched patients acutely admitted with a major depressive disorder. The patients are rated with a number of rating scales at admittance, day 5, after two weeks and three months. EEG and QEEG are taken three times the first week. MRI, drug screening and blood screening of medication-concentrations are taken.

ELIGIBILITY:
Inclusion Criteria:

* Acutely admitted psychiatric patients who have at different times the last 2 weeks filled criteria for at least two new DSM-4 Axis 1 psychiatric diagnoses. One of them has to be a depressive episode (MADRS>20)

Exclusion Criteria:

* Patients not speaking Norwegian or English.
* Patients not willing to participate.
* Patients with dementia or mental retardation to an extensive degree.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study and control groups both from a psychiatric acute ward. The patients are acutely admitted suffering from different types of depressive symptoms.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 1998-10; Primary Completion 2004-10 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
epilepsy or an other organic brain disorder | 1 week
  EEG and QEEG are taken three times in the first week

CONTACTS AND LOCATIONS:
Overall Officials: Olav M Linaker, Professor, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Østmarka Psychiatric Department, St. Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Vaaler AE, Morken G, Iversen VC, Kondziella D, Linaker OM. Acute Unstable Depressive Syndrome (AUDS) is associated more frequently with epilepsy than major depression. BMC Neurol. 2010 Jul 30;10:67. doi: 10.1186/1471-2377-10-67. PMID 20673344
- [Derived] Vaaler AE, Morken G, Linaker OM, Sand T, Kvistad KA, Brathen G. Symptoms of epilepsy and organic brain dysfunctions in patients with acute, brief depression combined with other fluctuating psychiatric symptoms: a controlled study from an acute psychiatric department. BMC Psychiatry. 2009 Sep 30;9:63. doi: 10.1186/1471-244X-9-63. PMID 19793395